CLINICAL TRIAL: NCT03734341
Title: A Telemonitoring Crossover Study Comparing a New Incremental Fixed Pressure Titration Modality Versus Auto-adjustable Titration for CPAP-naïve Obstructive Sleep Apnea Patients
Brief Title: Comparison of Two Telemonitoring Auto-titrating Modalities in OSA Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Mikel Azpiazu, Principal Investigator, Basque Health Service
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-37
Record Dates: First submitted 2018-11-06; First posted 2018-11-07 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Apnea; Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Sleep Disordered Breathing; Respiration; Sleep Disorder; Respiratory Tract Disease; Sleep Disorders, Intrinsic; Sleep Wake Disorders
Keywords: CPAP; Titration; Obstructive Sleep Apnea; Telemonitoring; Telemedicine
MeSH Terms: conditions — Apnea; Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Respiratory Aspiration; Sleep Wake Disorders; Respiratory Tract Diseases; Sleep Disorders, Intrinsic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EZ START Titration (Experimental): CPAP titration test performed with an auto CPAP device preset on incremental fixed pressure modality. If the titration pressure is achieved (in a 14-day maximum period) the device will be immediately and remotely preset in CPAP modality with EZ START pressure (if any) for a 14-day period to check the titration pressure performance in a short-time period.
  Afterwards, the device will be remotely preset on the next modality: auto-adjusting pressure (no wash-out period).
  Interventions: Device: EZ START Titration; Device: APAP Titration
- APAP Titration (Active Comparator): CPAP titration test performed with an auto CPAP device preset on auto-adjusting pressure modality. If the titration pressure is achieved (in a 14-day maximum period) the device will be immediately and remotely preset in CPAP modality with APAP pressure (if any) for a 14-day period to check the titration pressure performance in a short-time period.
  Afterwards, the device will be remotely preset on the next modality: incremental fixed pressure (no wash-out period).
  Interventions: Device: EZ START Titration; Device: APAP Titration

INTERVENTIONS:
Device: EZ START Titration — The auto CPAP device gradually increases air pressure night-by-night until the preset therapeutic pressure is reached.
  Pressure range: from 5 to 14 cmH2O. Ramp: 4cmH2O, 20 minutes. Mask: nasal (if no contraindication).
  Titration pressure: fixed pressure that reduces rAHI below 10, mask leak below 10% of the session, time session above 4 hours.
  Other Names: DreamStation auto CPAP; Philips Respironics; EncoreAnywhere
Device: APAP Titration — The auto CPAP device continuously adjusts the pressure in real time to the minimum pressure needed to maintain upper airway patency at any moment. Pressure range: 5 to 14 cm H2O. Ramp: 4cmH2O, 20 minutes. Mask: nasal (if no contraindication).
  Titration pressure: visual analysis pressure that reduces rAHI below 10 during 90% of the session, mask leak below 10% of the session, therapeutic session above 4 hours.
  Other Names: DreamStation auto CPAP; Philips Respironics; EncoreAnywhere

SUMMARY:
This study compares the titration pressures achieved through two auto-titrating modalities, a new incremental fixed pressure mode versus routine auto-adjusting pressure mode, in CPAP-naïve obstructive sleep apnea patients.

The aim of the study is to verify that this new modality achieves a lower titration pressure.

DETAILED DESCRIPTION:
In patients with obstructive sleep apnea (OSA) on CPAP treatment, a CPAP titration test is usually performed to achieve the optimal pressure to maintain upper airway patency, abolish obstructive respiratory events and reduce the occurrence of adverse events. This pressure is called titration pressure.

Until now, we used to perform, after an adaptation period, a single-night outpatient test with an automated device preset on auto-adjusting pressure modality (APAP).

The incremental fixed pressure modality (EZ START) was initially developed to ease patients into having a positive sleep therapy experience from the very beginning. This mode gradually increases air pressure night-by-night until the preset therapeutic pressure is reached. In each good therapy session, the device performs in fixed pressure overnight and we get a real residual apnea-hypopnea index (rAHI).

For this study, we will use the same device (DreamStation auto CPAP, Philips Respironics, Murrysville, PA, USA), a web-based system to telemonitor patient therapy (EncoreAnywhere) and perform for each individual patient the two modalities in a telemonitoring crossover randomized single-blind (patient) way.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* OSA diagnosis
* CPAP therapy indication

Exclusion Criteria:

* Previous CPAP therapy
* Severe COPD
* Respiratory insufficiency
* Obesity-hypoventilation syndrome
* Cardiac failure
* Recent cerebrovascular disease
* Central apnea, Cheyne Stokes or similar
* Important nasal insufficiency or malformation
* Previous pharyngeal surgery
* Shift work
* Psychosocial disability
* Refusal to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
Titration pressure | 14-day maximum period
  Titration pressure in any modality

SECONDARY OUTCOMES:
CPAP Adherence | 14-day period
  Adjusted adherence: days of use (%) * hours of use (mean)
CPAP Efficacy | 14-day period
  Residual AHI (mean) in the period

CONTACTS AND LOCATIONS:
Overall Officials: Mikel Azpiazu, MD, Principal Investigator — Basque Health Service
Locations (1):
- Hospital Universitario Araba, Vitoria-Gasteiz, Alava, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kushida CA, Chediak A, Berry RB, Brown LK, Gozal D, Iber C, Parthasarathy S, Quan SF, Rowley JA; Positive Airway Pressure Titration Task Force; American Academy of Sleep Medicine. Clinical guidelines for the manual titration of positive airway pressure in patients with obstructive sleep apnea. J Clin Sleep Med. 2008 Apr 15;4(2):157-71. PMID 18468315
- [Background] Masa JF, Jimenez A, Duran J, Capote F, Monasterio C, Mayos M, Teran J, Hernandez L, Barbe F, Maimo A, Rubio M, Montserrat JM. Alternative methods of titrating continuous positive airway pressure: a large multicenter study. Am J Respir Crit Care Med. 2004 Dec 1;170(11):1218-24. doi: 10.1164/rccm.200312-1787OC. Epub 2004 Jul 28. PMID 15282204
- [Background] McArdle N, Singh B, Murphy M, Gain KR, Maguire C, Mutch S, Hillman DR. Continuous positive airway pressure titration for obstructive sleep apnoea: automatic versus manual titration. Thorax. 2010 Jul;65(7):606-11. doi: 10.1136/thx.2009.116756. PMID 20627917
- [Background] Ahmed O, Parthasarathy S. APAP and Alternative Titration Methods. Sleep Med Clin. 2010 Sep 1;5(3):361-368. doi: 10.1016/j.jsmc.2010.05.010. PMID 20806054